CLINICAL TRIAL: NCT05201326
Title: An Open and Single-arm Prospective Clinical Study of the Safety and Efficacy of Irinotecan and Bevacizumab Combined With Re-radiotherapy in the Treatment of Recurrent Glioblastoma
Brief Title: Irinotecan And Bevacizumab Combined With Re-radiotherapy in Recurrent Glioblastoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, JIAYI CHEN, Chief of Department of Radiation Oncology, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJHGBMrRT
Record Dates: First submitted 2021-12-23; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): irinotecan + bevacizumab + Re-radiotherapy
  Interventions: Drug: Bevacizumab，Irinotecan and Re-radiotherapy

INTERVENTIONS:
Drug: Bevacizumab，Irinotecan and Re-radiotherapy — All patients with recurrent glioblastoma will accept irinotecan and bevacizumab combined with re-radiotherapy .

SUMMARY:
This is a phase I study to observe the safety and efficacy of irinotecan and bevacizumab combined with re-radiotherapy in the treatment of recurrent glioblastoma. The study will provide a higher level of clinical evidence-based evidence for the clinical treatment of recurrent GBM, and fill the guidelines for the treatment of recurrent GBM.

ELIGIBILITY:
Inclusion Criteria:

1. The initial diagnosis confirmed by histopathology is World Health Organization WHO grade 4 glioma;
2. Surgery, radiotherapy, chemotherapy, and adjuvant chemotherapy (Stupp plan) are performed after the initial diagnosis, and recurrence according to the evaluation of neurotumor response (RANO) criteria and/or confirmed by histopathology;
3. The expected survival period is ≥3 months;
4. Age between 18 and 70 years old;
5. KPS score (KPS) ≥ 70, able to take care of most of life, but occasionally need help from others;
6. There are measurable lesions on the T1 enhancement sequence of the head MRI;
7. Hematopoietic function: hemoglobin ≥90g/L, platelets ≥90×109/L, white blood cells ≥4×109/L (previous chronic anemia 80-90 g/L or previous low white blood cell level 3-4×109/L Or thrombocytopenia 80-90×109/L, but KPS 70-100 can be considered for admission) (The range of normal values can be fine-tuned due to the different standards of tertiary first-class hospitals);
8. Liver function: ALT and AST<1.5 times of high normal (ULN), bilirubin<1.5×ULN;
9. Sign the informed consent form;
10. Agree to participate in follow-up actions.

Exclusion Criteria:

1. Other invasive malignant tumors;
2. Re-irradiation after receiving recurrence in the past;
3. Recurrence more than 3 times or evidence that there is a subdural recurrence disease or a tumor with a maximum diameter of more than 6 cm;
4. Treat with vascular endothelial growth factor (VEGF) or VEGFR inhibitor or irinotecan in advance;
5. Pregnant or nursing mothers;
6. Participate in other tests after diagnosis of recurrence;
7. According to CTCAE5.0 standard classification of patients with bleeding above grade 3;
8. Symptomatic peripheral vascular disease;
9. Known allergy to bevacizumab or irinotecan;
10. Patients who are treated with anticoagulants or vitamin K antagonists such as warfarin, heparin or their analogs; under the premise that the prothrombin time international normalized ratio (INR) is ≤1.5, the use of small doses of Huafa for preventive purposes is allowed Farin (1 mg orally, once a day) or low-dose aspirin (do not exceed 100 mg per day);
11. Abnormal blood coagulation function, bleeding tendency (such as active peptic ulcer) or receiving thrombolysis or anticoagulation therapy;
12. Arterial/venous thrombotic events that occurred within 6 months before the first medication, such as cerebrovascular accidents (including temporary ischemic attacks), deep vein thrombosis and pulmonary embolism;
13. Urine routine test showed urine protein ≥++ and confirmed 24-hour urine protein quantification>1.0 g;
14. Long-term unhealed wounds or fractures;
15. Suffering from severe cardiovascular disease: myocardial ischemia or myocardial infarction above grade II, poor arrhythmia control (including men with QTc interval ≥450 ms, women ≥470 ms); according to NYHA standards, III to Grade IV insufficiency or color Doppler ultrasonography of the heart shows that the left ventricular ejection fraction (LVEF) is less than 50%;
16. Patients with hypertension who cannot be well controlled by a single antihypertensive drug treatment (systolic blood pressure> 140 mmHg, diastolic blood pressure> 90 mmHg), suffering from myocardial ischemia or myocardial infarction, arrhythmia (including QT room Period ≥440 ms) and degree I cardiac insufficiency;
17. History of organ transplantation;
18. According to the judgment of the researcher, a serious disease that endangers the safety of the patient or affects the completion of the study.
19. Poor overall health, even KPS<60;
20. Unable to understand the purpose of treatment or unwilling to sign the treatment consent form;
21. No capacity for civil conduct or limited capacity for civil conduct.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-12-22 (Actual); Primary Completion 2022-12-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
serious adverse events (SAE) | From baseline to 28 days after the end of treatment
  Clinical safety

SECONDARY OUTCOMES:
overall survival | From the beginning of treatment to death or the last follow-up, approximately 24 months
  the time between the date of enrollment of the patient and death from any cause
progression free survival | From the start of treatment to the date of disease progression or death, up to approximately 24 months
  The time between the patient's enrollment and any documented tumor progression or death from any cause.

OTHER OUTCOMES:
Quality of life score | Receive once every two months until you cannot tolerate toxicity or PD, up to about 24 months
  European Organization for Cancer Research and Treatment Quality of Life Questionnaire (EORTC QLQ-C30) Version 3.0 EORTC QLQ-C30 (Version 3.0) questionnaire for assessing quality of life.
Cognitive function | Receive once every two months until you cannot tolerate toxicity or PD, up to about 24 months
  The Mental State Test (MMSE, with a score ranging from 0 to 30) to assess cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayi Chen, MD, Study Director — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No